CLINICAL TRIAL: NCT04921553
Title: Real Word European Registry of NTRK Fusions and Other Rare Actionable Fusions (TRacKING)
Acronym: TRacKING
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Centre Leon Berard (Other)
Responsible Party: Sponsor
Other Study IDs: ET20000258 TRacKING
Record Dates: First submitted 2021-02-18; First posted 2021-06-10 (Actual); Last update posted 2021-08-02 (Actual); Status verified 2021-07

CONDITIONS: Cancer; Cancer Metastatic; NTRK Gene Fusion Overexpression; NTRK Family Gene Mutation; ATIC-ALK Fusion Protein Expression; ALK Fusion Protein Expression; BCR-FGFR1 Fusion Protein Expression; ROS1 Gene Translocation; COL1A1-PDGFB Fusion Protein Expression; RET Gene Translocation; Gene Fusion; ROS Gene Translocation; BRAF Gene Rearrangement; FGFR2 Gene Translocation; FGFR3 Gene Translocation; NTRK1 Gene Translocation
Keywords: actionnable fusion; cancer; registry; European reference network
MeSH Terms: conditions — Neoplasms; Neoplasm Metastasis | interventions — Data Collection

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 2 Years
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Data collection and quality of life questionnaire — * Data collection from the medical file
  * Quality of life questionnaire (QLQC30) at inclusion, at each change of treatment and then every 6 months

SUMMARY:
This registry will make it possible to describe real life management of patients with rare actionable fusions and to better understand these cancers. In addition of clinical data from the medical files, a quality of life questionnaire (QLQ-C30) will be complete at inclusion, at each new treatment and then every 6 months. The patients will be followed for a period of at least 2 years after the inclusion.

This TRacKING registry is a European collaborative tool to improve the management of patients with actionable fusions, by sharing of data from rare tumor indications.

DETAILED DESCRIPTION:
1. Administrative opening of the center
2. Routine identification of a patients harboring a rare actionable fusion
3. Patient's inclusion

   * Signature of written informed consent,
   * Declaration by the physician to the coordinating center (using the "Physician declaration" form)
   * Completion of the QLQ-C30 questionnaire (at inclusion, at each new treatment and then every 6 months).
4. Collection of retrospective and prospective data into the e-CRF by a local CRA using patients' medical files.

ELIGIBILITY:
Inclusion Criteria:

* Patient with histologically-confirmed cancer
* Patient harboring a rare actionable fusion (see Appendix 1),
* Availability of clinical and demographic data, information on treatment and clinical outcome.
* Adult, ≥18 years old,
* Patient should understand, sign and date the written voluntary informed consent form.

Exclusion Criteria:

-

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Patient with histologically-confirmed cancer that harboring a rare actionnable fusion, treated in a European center
Sampling Method: Non-Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2021-06-22 (Actual); Primary Completion 2025-06 (Estimated); Study Completion 2025-06 (Estimated)

PRIMARY OUTCOMES:
Overall Survival | 2 years
  To describe the survival rate of patients with solid cancers harboring a NTRK fusion or other rare actionable fusion in real-life practice, according to overall survival (OS)

SECONDARY OUTCOMES:
Management of patient with actionable fusion | up to 48 months
  Treatment scheme : number of line and type of treatments
Time to relapse | up to 48 months
Progression Free Survival (PFS) | after 6, 12 and 24 months
Incidence of long-term responders | up to 48 months
  long term responders =: > 24 months
Quality of life of patient | After 6, 12, 18, 24, 30, 36, 42, 48 months
  To evaluate patient-reported outcomes concerning individual QoL according to QLQ-C30 (EORTC Quality of Life questionnaires)
Time to relapse for fusion-targeting treatments | up to 48 months
Overall survival for patient treated by fusion-targeting treatments | 2 years
PFS for patient treated by fusion-targeting treatments | After 6, 12, 24 months of treatment by fusion targeting treatments
  Progression free survival
Incidence of long-term responders for patient treated by fusion-targeting treatments | up to 48 months
  > 24 months
Quality of life of patient treated by fusion-targeting treatments | After 6, 12, 18, 24, 30, 36, 42, 48 months of fusion-targeting treatments
  using QLQC30 (EORTC Quality of Life questionnaires)
Safety : Nature of adverse reaction (for treatment targeting a fusion) | up to 48 months
  Using Common Terminology Criteria for Adverse Events (CTCAE) V5.0.
Safety : Frequency of adverse reaction (for treatment targeting a fusion) | up to 48 months
  Using Common Terminology Criteria for Adverse Events (CTCAE) V5.0.
Safety : Severity of adverse reaction (for treatment targeting a fusion) | up to 48 months
  Using Common Terminology Criteria for Adverse Events (CTCAE) V5.0.

CONTACTS AND LOCATIONS:
Overall Officials: Jean-Yves BLAY, Pr, Principal Investigator — Centre Leon Berard
Locations (41):
- Austria (2):
  - University Hospital Graz, Graz
  - Medical University of Vienna, Vienna
- Masaryk Memorial Cancer Institute (Masarykuv Onkologicky Ustav), Brno, Czechia
- Aarhus University Hospital, Aarhus, Denmark
- France (14):
  - Chu Jean Minjoz, Besançon
  - Institut Bergonie, Bordeaux
  - Centre Georges Francois Leclerc, Dijon
  - Centre Oscar Lambret, Lille
  - Chu Dupuytren, Limoges
  - Centre Léon Bérard, Lyon
  - Assistance Publique Hopitaux de Marseille (AP-HM), Marseille
  - Centre Antoine Lacassagne, Nice
  - Institut Curie, Paris
  - Aphp - Hopital de La Pitie Salpetriere, Paris
  - Aphp - Hopital Cohin, Paris
  - Aphp - Hopital Tenon, Paris
  - Centre Henri Becquerel, Rouen
  - Institut Claudius Regaud, Toulouse
- Germany (11):
  - "Hämato-Onkologischer Studienkreis MVZ am Klinikum Aschaffenburg / Onkologie", Aschaffenburg
  - Charité - Universitätsmedizin Berlin, Berlin
  - "Klinik für Innere Medizin III, Hämatologie, Onkologie Klinikum Chemnitz", Chemnitz
  - "Medizinische Klinik 1- Gastroenterologie, Hepatologie, Pneumologie Universitätsklinikum Frankfurt", Frankfurt am Main
  - "Hämatologisch-onkologische Ambulanz Universitätsklinikum Halle", Halle
  - "Klinik für Gastroenterologie, Hepatologie und Infekt Universitätsklinikum Magdeburg", Magdeburg
  - Mannheim University Medical Center (UniversitatsMedizin Mannheim), Mannheim
  - "Medizinische Klinik und Poliklinik III LMU - Klinikum der Universität München", München
  - "Klinik für Innere Medizin III, Hämatologie, Onkologie Südharzklinikum", Nordhausen
  - Universitätsklinikum Tübingen Medizinische Universitätsklinik;, Tübingen
  - University Hospital Würzburg (UniversitätsKlinikum Würzburg), Würzburg
- Italy (6):
  - Azienda Ospedaliera - Universitaria - Policlinico S Orsola-Malpighi Univertsita di Bologna, Bologna
  - Istituto Scientifico Romagnolo per lo Studio e la Cura dei Tumori, Meldola
  - Fondazione IRCCS Istituto Neurologico Carlo Besta, Milan
  - IRCCS Ospedale San Raffale, Milan
  - CRTR-AOU Federico II, Napoli
  - Azienda Ospedaliero - Universitaria Cita della Salute e della Scienza di Torino, Torino
- Leiden University Medical Center, Leiden, Netherlands
- Maria Sklodowska Curie National Research Institute of Oncology, Warsaw, Poland
- Institute of Oncology of Ljubljana, Ljubljana, Slovenia
- Complejo Hospitalario regional Virgen del Rocio, Seville, Spain
- United Kingdom (2):
  - The Royal Marsden NHS Foundation Trust, London
  - University College London NHS Foundation Trust, London

IPD SHARING:
Plan to Share IPD: No